CLINICAL TRIAL: NCT00670293
Title: Imaging of Dopamine Systems in Anorexia Nervosa
Brief Title: Changes in Dopamine Levels Before and After Weight Restoration in People With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5700; R01MH079397 (NIH)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2015-08

CONDITIONS: Eating Disorders
Keywords: Anorexia Nervosa; PET Imaging; Dopamine
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Methylphenidate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with anorexia nervosa: Underweight participants with anorexia nervosa who will restore normal weight levels after inpatient treatment will undergo Positron Emission Tomography (PET) using [11C]raclopride as well as MRI
  Interventions: Radiation: Positron Emission Tomography (PET) using [11C]raclopride; Drug: Methylphenidate; Procedure: Magnetic Resonance Imaging (MRI) scan
- Healthy weight controls: Participants who are healthy controls will undergo Positron Emission Tomography (PET) using [11C]raclopride as well as MRI
  Interventions: Radiation: Positron Emission Tomography (PET) using [11C]raclopride; Drug: Methylphenidate; Procedure: Magnetic Resonance Imaging (MRI) scan

INTERVENTIONS:
Radiation: Positron Emission Tomography (PET) using [11C]raclopride — Participants with AN will undergo three PET scans at two separate time points. The first scan will occur when participants are underweight (but not less than 75% ideal body weight), and the second and third scans will occur 2 to 4 weeks after participants have accomplished weight restoration. Healthy participants will have two PET scans at a single timepoint.
Drug: Methylphenidate — The second PET scan for healthy participants and third PET scan for participants with AN will be performed after administration of 60 mg of methylphenidate, a psychostimulant that allows for accumulation of dopamine (DA) extraneuronally.
Procedure: Magnetic Resonance Imaging (MRI) scan — Participants with AN will undergo two MRI scans, and healthy participants will undergo one MRI scan. The scans will be conducted in conjunction with the PET scans.

SUMMARY:
This study will use positron emission tomography imaging to investigate changes in dopamine systems in people with anorexia nervosa before and after weight restoration.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a disordered eating disease characterized by a persistent pursuit of thinness, intense fear of weight gain, distorted body image, and obsessive eating habits. People with AN are at high risk for certain health problems, such as depression, osteoporosis, substance abuse, and cardiovascular and neurological complications. Current treatments for AN include different forms of psychotherapy and medications, but the success of these treatments is highly variable among people with AN. A better pathophysiologic understanding of AN is needed in order to develop novel therapeutic strategies for preventing and treating the disorder. Current research is targeting dopamine (DA), a neurotransmitter that is released in response to pleasurable stimuli, such as food and drugs. Animal studies have found that chronic food restriction may alter functioning of the DA system by reducing DA response to food and drug stimuli. A better understanding of the effects of disordered eating on the DA systems of people with AN may provide insight into the development of new and improved treatments for people with AN. This study will use positron emission tomography (PET) imaging to investigate changes in DA systems in people with AN before and after both weight restoration and administration of methylphenidate, a psychostimulant medication. The study will also use PET imaging to compare DA systems of people with AN with DA systems of people who are healthy.

This study will involve both healthy participants and participants with AN. Study participation for healthy participants will include two PET scans and one magnetic resonance imaging (MRI) scan, which, if the participants prefer, can all be completed in one study visit. Study participation for participants with AN will include three PET and two MRI scans. The first PET and MRI scans will be performed upon entry into the hospital as an inpatient. The remaining scans will be conducted 2 to 4 weeks after participants have accomplished weight restoration.

Including preparation, each MRI study will last about 45 minutes and each PET study will last about 3 hours. For each MRI study, participants will be asked to lie on their backs for 15 minutes in the MRI scanner. For each PET study, participants will first be injected with a dose of [11C]raclopride, a radioactive drug used in brain imaging, and will then lie on their backs for 30 minutes in the PET scanner.

One hour before the second PET scan for healthy participants and the third PET scan for participants with AN, participants will receive an oral dose of methylphenidate. During these scans, participants will also undergo blood pressure monitoring and an electrocardiogram (EKG). Once participants no longer feel the effects of the methylphenidate and their vital signs have returned to normal, they will be discharged from the medical center and study participation will be complete.

ELIGIBILITY:
Inclusion Criteria:

Participants with AN:

* Meets DSM-IV criteria for AN or ED-NOS (meets criteria for AN except amenorrhea)
* Sufficiently medically and psychiatrically stable to leave inpatient unit, as assessed by clinical team

Healthy control participants:

* No current or past psychiatric illness
* Between 80% and 120% of ideal body weight

Exclusion Criteria:

All participants:

* Current use of psychotropic medication such as antipsychotics or antidepressants
* Pregnant or breastfeeding
* History of a substance use disorder
* Significant medical illness
* High blood pressure (resting systolic blood pressure greater than 140 mmHg and diastolic blood pressure greater than 90 mmHg)
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV-TR
* Metal implants or paramagnetic objects contained within the body that may interfere with the MRI scan, as determined in consultation with a neuroradiologist and according to specified reference book guidelines
* Exposed to radiation in the workplace or has had a nuclear medicine procedure during the 1 year before study entry
* Previous adverse reaction to psychostimulants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include people with anorexia nervosa seeking inpatient treatment or already receiving inpatient treatment and people who will act as healthy control participants.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Dopamine receptor binding potential | Measured at baseline and after healthy weight restoration

CONTACTS AND LOCATIONS:
Overall Officials: Allegra Broft, MD, Principal Investigator — The New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States